CLINICAL TRIAL: NCT03321851
Title: An Open Label, Interventional, Clinical Performance and Validation Study to Demonstrate the Clinical Accuracy of of the V-Sensor in the Healthy Adult Population; Single Site in Switzerland
Brief Title: V-Sensors for Vitals: Assessment of the Accuracy of a Vital Sign Sensor Mounted on a Smartphone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Léman Micro Devices SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LMD-CT-002
Record Dates: First submitted 2017-10-12; First posted 2017-10-26 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2017-10

CONDITIONS: Clinical Accuracy of Vital Sign Pressure Sensor

STUDY DESIGN:
Intervention Model Description: Each participant tests two equivalent vital sign sensors (devices under test) mounted on two different smartphones, one after another to assess accuracy of the device compared to equivalent reference devices.
Masking Description: Vital sign results obtained by the device under study are not displayed on phone screen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-Sensor Device User (Other): This diagnostic medical device is designed to detect the user's 5 vital signs. Each user tests two sensors, each sensor is mounted on a smartphone. Each vital sign is compared to an equivalent reference device obtained by the healthcare provider.
  Interventions: Device: V-sensor device user

INTERVENTIONS:
Device: V-sensor device user — Participants use device to detect the 5 vital signs (Blood Pressure, Pulse, Respiration, SpO2, Temperature).

SUMMARY:
This trial seeks to demonstrate clinical accuracy and safety of the integrated V-Sensor when used by the general, healthy adult population interested in measuring their vital signs outside of the clinical setting.

DETAILED DESCRIPTION:
The five vital signs are blood pressure, pulse, respiration, SpO2, and temperature. The user tests two devices mounted on two smartphones.

* Temperature: Each user will use the V-sensor mounted on a smartphone to obtain his/her temperature interfaced with a temperature specific 'app'. Before and after the the temperature is obtained using the V-Sensor, the temperature will be obtained using an equivalent thermometer.
* Blood Pressure: Each user will test his/her blood pressure using the two sensors mounted on the two phones interfaced with a blood pressure specific 'app'. Before and after each measurement, a reference measurement using a mercury sphygmomanometer will be taken.
* Pulse, Respiration, SpO2: Each user will test his/her pulse, respiration, and SpO2 using 2 V-sensors mounted on two separate smartphones interfaced with a Pulse, Respiration, and SpO2 'app'. Before and after each measurement, a reference measurement using equivalent reference devices will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* 18 and 80 years old
* no history or risk for developing lymphedema
* no arteriovenous fistula in the right arm
* no right limb amputation up to and including the right index finger
* ability to obtain 3 readings from the device during the screening/training session.

Exclusion Criteria:

* history of arrhythmia
* arteriovenous fistula in the right arm
* lymphedema or high risk for developing lymphedema in the right arm
* inability to follow the procedures of the study
* inability to hold the study device as instructed
* inability to obtain 3 readings from the study device during the screening session
* previous enrolment into the current study
* enrolment of the Investigator or Sponsor, his/her family members, employees and other dependent persons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure accuracy to the reference device within the ranges specified by the ISO standard 81060-2 | 4 months
  For systolic and diastolic blood pressures, the mean error of determination of the individual paired determinations of the sphygmomanometer-under-test and the reference sphygmomanometer (Standby Baumanometer) for all participants shall not be greater than 8.0mmHg.
Pulse Rate accuracy to the reference device within the ranges specified by the ISO 80601-2-61 | 4 months
  Pulse rate accuracy shall be stated as the root-mean-square (rms) difference between paired pulse rate data recorded with the pulse oximeter equipment and with the Nellcor N-PA reference device.
Blood Oxygen accuracy to the reference device within the ranges specified by the ISO 80601-2-61. | 4 months
  The SpO2 accuracy shall be stated as a root-mean-square (rms) difference of less than or equal to 4.0% SpO2 over the range of 70% to 100% SaO2
Respiration rate accuracy | 4 months
  Respiration rate accuracy shall be stated as the root-mean-square (rms) difference between paired respiratory rate data with the Passport Respiration Rate Sensor PS-2133 reference method; target range +/- 10% of participant's respiratory rate
Temperature accuracy to the reference device with the ranges specified by the ISO 80601-2-56 & ATSM 1965 Standard. | 4 months
  Temperature accuracy shall be stated as the root-mean-square (rms) difference between paired temperatures data recorded with the Exergen Temporal Scanner thermometer. LMD's target is a clinical bias <= 3.0°C and a clinical repeatability <= 3.0°C.

SECONDARY OUTCOMES:
No serious adverse device effects are reported. | 4 months
  Zero serious adverse device effects are reported.

CONTACTS AND LOCATIONS:
Overall Officials: Chris J Elliott, PhD, Study Director — Leman Micro-Device

IPD SHARING:
Plan to Share IPD: No